CLINICAL TRIAL: NCT03328897
Title: A Phase III Study to Evaluate the Efficacy and Safety of Xolair® (Omalizumab) in Chinese Patients With Chronic Spontaneous Urticaria (CSU) Who Remain Symptomatic Despite Antihistamine Treatment
Brief Title: Study of Efficacy and Safety of Xolair® (Omalizumab) in Chinese Patients With Chronic Spontaneous Urticaria
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CIGE025E2305
Record Dates: First submitted 2017-03-13; First posted 2017-11-01 (Actual); Results first posted 2020-11-04 (Actual); Last update posted 2020-11-04 (Actual); Status verified 2020-10

CONDITIONS: Chronic Spontaneous Urticaria
Keywords: Chronic spontaneous urticaria; ISS7; UAS7; omalizumab; China
MeSH Terms: conditions — Chronic Urticaria | interventions — Omalizumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Omalizumab 300mg (Experimental): patients received a dose of omalizumab 300 mg which consisted of two injections of omalizumab 150 mg vials every 4 weeks (Day 1, Week 4 and Week 8)
  Interventions: Drug: Omalizumab
- Omalizumab 150mg (Experimental): patients received a dose of omalizumab 150 mg which consisted of one injection of omalizumab 150 mg vial and one injection of placebo 150 mg vial every 4 weeks (Day 1, Week 4 and Week 8)
  Interventions: Drug: Omalizumab
- Placebo (Placebo Comparator): patients received placebo which consisted of two injections of placebo 150 mg vials every 4 weeks (Day 1, Week 4 and Week 8)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Omalizumab — injection of 150mg or 300 mg
  Other Names: IGE025
  Arms: Omalizumab 150mg; Omalizumab 300mg
Drug: Placebo — Injection of placebo
  Arms: Placebo

SUMMARY:
The purpose of this study was to demonstrate the efficacy and safety of omalizumab, compared with placebo, as an add-on to H1 antihistamines (H1AH) therapy in adult patients suffering from Chronic Spontaneous Urticaria (CSU) who remained symptomatic despite H1AH therapy.

DETAILED DESCRIPTION:
This was a randomized, multicenteric, double-blinded, placebo-controlled, parallel-group study to evaluate the efficacy and safety of omalizumab as an add-on therapy for the treatment of patients of refractory CSU who remained symptomatic despite approved-dosed H1AH treatment.

The study consisted of three distinct epochs over 24 weeks: Screening epoch (Day -28 to Day -1), Randomized treatment epoch (Day 1 to Week 12) and Post-treatment follow-up epoch (Week 12 to Week 20). Patients were randomized into three treatment groups (omalizumab 300 mg s.c. omalizumab 150 mg s.c. and placebo) in a 2:2:1 ratio, stratified by latent tuberculosis (TB) status at Baseline (Yes/No).

On Day 1, eligible patients were randomly assigned to receive omalizumab (150 mg or 300 mg) or placebo by subcutaneous (s.c.) injection every 4 weeks (on Day 1, Week 4, and Week 8) during the 12-week double-blind randomized-treatment epoch. Patients visited the study center at 4-week intervals. Patients were instructed to stay on the same CSU H1AH treatment at stable dose that they were using during the pre-randomization period during the randomized treatment epoch. They were allowed to use diphenhydramine as rescue medication during all epochs. The last dose of the study drug during the randomized-treatment epoch was administered at Week 8 study visit, however, the last assessment was done at Week 12.

After the completion of the 12-week randomized-treatment epoch, all patients entered an 8-week post-treatment follow-up epoch.

ELIGIBILITY:
Main Inclusion Criteria:

* Symptomatic CSU patients with CSU diagnosis for at least 6 months.
* Patients must have been on an approved dose of an H1AH for CSU for at least the 3 consecutive days immediately prior to the Day -14 screening visit
* Patients must have documented current use on the day of the initial screening visit

Main Exclusion Criteria

* Clearly defined underlying etiology for chronic urticarias other than CSU (main manifestation being physical urticaria)
* Other skin disease associated with itch Urticarial vasculitis, urticaria pigmentosa, erythema multiforme, mastocytosis, hereditary or acquired angioedema, lymphoma, leukemia, or generalized cancer

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 418 (Actual)
Dates: Start 2017-04-26 (Actual); Primary Completion 2019-07-23 (Actual); Study Completion 2019-09-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (19):
- China (19):
  - Novartis Investigative Site, Beijing, Beijing Municipality
  - Novartis Investigative Site, Fuzhou, Fujian
  - Novartis Investigative Site, Guangzhou, Guangdong
  - Novartis Investigative Site, Nanning, Guangxi
  - Novartis Investigative Site, Harbin, Heilongjiang
  - Novartis Investigative Site, Wuhan, Hubei
  - Novartis Investigative Site, Changsha, Hunan
  - Novartis Investigative Site, Nanjing, Jiangsu
  - Novartis Investigative Site, Suzhou, Jiangsu
  - Novartis Investigative Site, Wuxi, Jiangsu
  - Novartis Investigative Site, Shenyang, Liaoning
  - Novartis Investigative Site, Chengdu, Sichuan
  - Novartis Investigative Site, Ürümqi, Xinjiang
  - Novartis Investigative Site, Hangzhou, Zhejiang
  - Novartis Investigative Site, Beijing
  - Novartis Investigative Site, Chongqing
  - Novartis Investigative Site, Guangzhou
  - Novartis Investigative Site, Nanjing
  - Novartis Investigative Site, Shanghai

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com

REFERENCES:
- [Derived] Bi XD, Lu BZ, Pan XX, Liu S, Wang JY. Adjunct therapy with probiotics for chronic urticaria in children: randomised placebo-controlled trial. Allergy Asthma Clin Immunol. 2021 Apr 17;17(1):39. doi: 10.1186/s13223-021-00544-3. PMID 33865434

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were recruited from 27 sites across China.
Pre-assignment Details: Patients were randomized into three treatment groups (omalizumab 300 mg s.c., omalizumab 150 mg s.c. and placebo) in a 2:2:1 ratio.
Period: Randomized-treatment Epoch
Arm/Group | Omalizumab 300mg | Omalizumab 150mg | Placebo
Started (Randomized) | 168 | 167 | 83
Full Analysis Set (FAS) (includes all randomized patients who took at least one dose of study medication.) | 167 | 167 | 83
Completed (Completed randomized-treatment epoch) | 152 | 162 | 81
Not Completed | 16 | 5 | 2
Not completed — Adverse Event | 4 | 1 | 1
Not completed — Lost to Follow-up | 0 | 1 | 0
Not completed — Pregnancy | 3 | 0 | 0
Not completed — Patient/guardian decision | 8 | 3 | 1
Not completed — Lack of Efficacy | 1 | 0 | 0
Period: Follow-up Epoch
Arm/Group | Omalizumab 300mg | Omalizumab 150mg | Placebo
Started (Entered follow-up epoch) | 161 | 163 | 81
Completed (Completed follow-up epoch) | 153 | 160 | 79
Not Completed | 8 | 3 | 2
Not completed — Adverse Event | 4 | 0 | 1
Not completed — Lack of Efficacy | 1 | 1 | 1
Not completed — Lost to Follow-up | 0 | 1 | 0
Not completed — Pregnancy | 1 | 0 | 0
Not completed — Patient/guardian decision | 2 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Omalizumab 300mg | Omalizumab 150mg | Placebo | Total
Number analyzed (Participants) | 168 | 167 | 83 | 418
Age, Continuous [Mean (Standard Deviation); unit: years] | 40.4 (12.29) | 38.8 (12.18) | 42.8 (12.32) | 40.2 (12.31)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 115 | 108 | 53 | 276
  Male | 53 | 59 | 30 | 142
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: Asian | 168 | 167 | 83 | 418
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Ethnicity: Chinese | 168 | 167 | 83 | 418

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline of the Itch Severity Score (ISS7) Score After 12 Weeks of Treatment
Description: The severity of the itch was recorded by the patient twice daily in their eDiary, on a scale of 0 (none) to 3 (intense/severe). Baseline ISS7 was calculated 7 days prior to the first treatment date. A weekly score (ISS7) was derived by adding up the average daily scores of the seven days preceding the visit. The possible range of the weekly score was therefore 0 to 21, where 0 is the best score and 21 is the worst score. The complete itch response was defined as ISS7 = 0.
  Itch (Pruritus) Severity Score Scale:
  0 = None
  1. = Mild (minimal awareness, easily tolerated)
  2. = Moderate (definite awareness, bothersome but tolerable)
  3. = Severe (difficult to tolerate)
Time Frame: Baseline, Week 12
Population: Full Analysis Set
Measure: Least Squares Mean (Standard Error); unit: Score on a scale
Arm/Group | Omalizumab 300mg | Omalizumab 150mg | Placebo
Number analyzed (Participants) | 167 | 167 | 83
Score on a scale | -10.11 (0.430) | -9.66 (0.424) | -5.87 (0.604)
Statistical Analysis 1: Comparison: Omalizumab 300mg vs Placebo; Test type: Superiority; p < 0.001, Mixed Model with Repeated Measures(MMRM); Mean Difference (Net) = -4.23, 95% CI 2-sided [-5.70 to -2.77], Standard Error of Mean 0.746
Statistical Analysis 2: Comparison: Omalizumab 150mg vs Placebo; Test type: Superiority; p < 0.001, Mixed Model with Repeated Measures(MMRM); Mean Difference (Net) = -3.79, 95% CI 2-sided [-5.24 to -2.33], Standard Error of Mean 0.738

2. Secondary Outcome: Change From Baseline of Urticaria Activity Score (UAS7) After 12 Weeks of Treatment
Description: UAS7 is the sum of the HSS7 and the ISS7 scores. The possible range of the weekly UAS7 score is 0 to 42. A higher urticaria activity score indicates more severe symptoms. A negative change score from baseline indicates improvement.
Time Frame: Baseline, Week 12
Population: Full Analysis Set
Measure: Least Squares Mean (Standard Error); unit: Score on a scale
Arm/Group | Omalizumab 300mg | Omalizumab 150mg | Placebo
Number analyzed (Participants) | 167 | 167 | 83
Score on a scale | -21.82 (0.895) | -20.74 (0.882) | -11.62 (1.258)
Statistical Analysis 1: Comparison: Omalizumab 300mg vs Placebo; Test type: Superiority; p < 0.001, Mixed Model with Repeated Measures(MMRM); Mean Difference (Net) = -10.19, 95% CI 2-sided [-13.25 to -7.14], Standard Error of Mean 1.555
Statistical Analysis 2: Comparison: Omalizumab 150mg vs Placebo; Test type: Superiority; p < 0.001, Mixed Model with Repeated Measures(MMRM); Mean Difference (Net) = -9.12, 95% CI 2-sided [-12.14 to -6.10], Standard Error of Mean 1.535

3. Secondary Outcome: Change From Baseline of Number of Hives Score (NHS7) After 12 Weeks of Treatment
Description: Hives Severity Score (HSS), defined by number of hives, were recorded by the patient twice daily in their eDiary, on a scale of 0 (none) to 3 (intense/severe). A weekly number of hives score (NHS7) was derived by adding up the average daily scores of the seven days preceding the visit. The possible range of the weekly score was therefore 0 to 21. The complete hives response was defined as NHS7 = 0.
  Hives Severity Score scale:
  0 - None
  * Mild (1-6 hives/12 hours)
  * Moderate (7-12 hives/12 hours)
  * Severe (>12 hives/12 hours)
Time Frame: Baseline, Week 12
Population: Full analysis set
Measure: Least Squares Mean (Standard Error); unit: Score on a scale
Arm/Group | Omalizumab 300mg | Omalizumab 150mg | Placebo
Number analyzed (Participants) | 167 | 167 | 83
Score on a scale | -11.68 (0.492) | -11.11 (0.485) | -5.76 (0.690)
Statistical Analysis 1: Comparison: Omalizumab 300mg vs Placebo; Test type: Superiority; p < 0.001, Mixed Model with Repeated Measures(MMRM); Mean Difference (Net) = -5.92, 95% CI 2-sided [-7.59 to -4.24], Standard Error of Mean 0.853
Statistical Analysis 2: Comparison: Omalizumab 150mg vs Placebo; Test type: Superiority; p < 0.001, Mixed Model with Repeated Measures(MMRM); Mean Difference (Net) = -5.35, 95% CI 2-sided [-7.00 to -3.69], Standard Error of Mean 0.842

4. Secondary Outcome: Percentage of Patients With UAS7≤6 at Week 12
Description: UAS7 is the sum of the HSS7 and the ISS7 scores. The possible range of the weekly UAS7 score is 0 to 42. A higher urticaria activity score indicates more severe symptoms. A negative change score from baseline indicates improvement. Week 12 responders were defined as patients who achieved an absolute UAS7 ≤ 6 at Week 12. A patient with missing data at Week 12 was imputed as a responder if the patient was a responder at Week 10 and Week 11, otherwise as a non-responder.
Time Frame: Week 12
Population: Full analysis set
Measure: Count of Participants; unit: Participants
Arm/Group | Omalizumab 300mg | Omalizumab 150mg | Placebo
Number analyzed (Participants) | 167 | 167 | 83
Participants | 81 | 79 | 9
Statistical Analysis 1: Comparison: Omalizumab 300mg vs Placebo; Test type: Superiority; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 7.02, 95% CI 2-sided [3.27 to 15.06]
Statistical Analysis 2: Comparison: Omalizumab 150mg vs Placebo; Test type: Superiority; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 7.03, 95% CI 2-sided [3.29 to 15.06]

5. Secondary Outcome: Percentage of Complete Responders (UAS7 = 0) at Week 12
Description: UAS7 is the sum of the HSS7 and the ISS7 scores. The possible range of the weekly UAS7 score is 0 to 42. A higher urticaria activity score indicates more severe symptoms. A negative change score from baseline indicates improvement. Complete responders are defined as participants who achieved UAS7 = 0.
Time Frame: Week 12
Population: Full analysis set
Measure: Count of Participants; unit: Participants
Arm/Group | Omalizumab 300mg | Omalizumab 150mg | Placebo
Number analyzed (Participants) | 167 | 167 | 83
Participants | 62 | 39 | 4
Statistical Analysis 1: Comparison: Omalizumab 300mg vs Placebo; Test type: Superiority; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 11.21, 95% CI 2-sided [3.88 to 32.37]
Statistical Analysis 2: Comparison: Omalizumab 150mg vs Placebo; Test type: Superiority; p = 0.001, Regression, Logistic; Odds Ratio (OR) = 5.88, 95% CI 2-sided [2.01 to 17.17]

6. Secondary Outcome: Percentage of Patients With ISS7 Minimally Important Difference (MID) at Week 12
Description: The severity of the itch was recorded by the patient twice daily in their eDiary, on a scale of 0 (none) to 3 (intense/severe). Baseline ISS7 was calculated 7 days prior to the first treatment date. A weekly score (ISS7) was derived by adding up the average daily scores of the seven days preceding the visit. The possible range of the weekly score was therefore 0 to 21, where 0 is the best score and 21 is the worst score. The complete itch response was defined as ISS7 = 0.
  Itch (Pruritus) Severity Score Scale:
  0 = None
  1. = Mild (minimal awareness, easily tolerated)
  2. = Moderate (definite awareness, bothersome but tolerable)
  3. = Severe (difficult to tolerate)
  The ISS7 MID response was defined as a reduction from Baseline in ISS7 of ≥ 5 points.
Time Frame: Week 12
Population: Full analysis set
Measure: Count of Participants; unit: Participants
Arm/Group | Omalizumab 300mg | Omalizumab 150mg | Placebo
Number analyzed (Participants) | 167 | 167 | 83
Participants | 125 | 125 | 49
Statistical Analysis 1: Comparison: Omalizumab 300mg vs Placebo; Test type: Superiority; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 2.73, 95% CI 2-sided [1.51 to 4.95]
Statistical Analysis 2: Comparison: Omalizumab 150mg vs Placebo; Test type: Superiority; p = 0.002, Regression, Logistic; Odds Ratio (OR) = 2.53, 95% CI 2-sided [1.41 to 4.56]

7. Secondary Outcome: Change From Baseline of Dermatology Life Quality Index (DLQI) Score After 12 Weeks of Treatment
Description: Dermatology life quality index (DLQI) is a 10-item dermatology- specific health-related quality of life measure. Patients rated their dermatology symptoms as well as the impact of their skin condition on various aspects of their lives. An overall score was calculated as well as separate scores for the following domains: symptoms and feelings, daily activities, leisure, work and school, personal relationships, treatment. Each domain had 4 response categories ranging from 0 (not at all) to 3 (very much). "Not relevant" is a valid score also and is scored as 0. The DLQI total score is a sum of all 10 responses. Scores range from 0 to 30 with higher scores indicating greater health-related quality of life impairment.
Time Frame: Week 12
Population: Full analysis set
Measure: Least Squares Mean (Standard Error); unit: Score on a scale
Arm/Group | Omalizumab 300mg | Omalizumab 150mg | Placebo
Number analyzed (Participants) | 167 | 167 | 83
Score on a scale | -10.4 (0.50) | -9.9 (0.49) | -6.5 (0.69)
Statistical Analysis 1: Comparison: Omalizumab 300mg vs Placebo; Test type: Superiority; p < 0.001, Mixed Model with Repeated Measures(MMRM); Mean Difference (Net) = -4.0, 95% CI 2-sided [-5.7 to -2.3], Standard Error of Mean 0.85
Statistical Analysis 2: Comparison: Omalizumab 150mg vs Placebo; Test type: Superiority; p < 0.001, Mixed Model with Repeated Measures(MMRM); Mean Difference (Net) = -3.5, 95% CI 2-sided [-5.1 to -1.8], Standard Error of Mean 0.85

8. Secondary Outcome: Time to ISS7 MID Response by Week 12
Description: The ISS7 MID response was defined as a reduction from Baseline in ISS7 of ≥ 5 points. Time to ISS7 MID response was the time (in weeks) from the date of the first dose to the date where ISS7 MID response was first achieved during Week 1 to Week 12.
Time Frame: 12 weeks
Population: Full analysis set
Measure: Count of Participants; unit: Participants
Arm/Group | Omalizumab 300mg | Omalizumab 150mg | Placebo
Number analyzed (Participants) | 167 | 167 | 83
Participants
  First Response: >0 to <=4 weeks | 114 | 109 | 42
  First Response: >4 to <=8 weeks | 18 | 25 | 10
  First Response: >8 to <=12 weeks | 10 | 10 | 7
  No response | 25 | 23 | 24
Statistical Analysis 1: Comparison: Omalizumab 300mg vs Placebo; Test type: Superiority; p < 0.001, Regression, Cox; Hazard Ratio (HR) = 1.71, 95% CI 2-sided [1.25 to 2.33]
Statistical Analysis 2: Comparison: Omalizumab 150mg vs Placebo; Test type: Superiority; p = 0.001, Regression, Cox; Hazard Ratio (HR) = 1.66, 95% CI 2-sided [1.22 to 2.25]

ADVERSE EVENTS:
Time Frame: Adverse events were collected from first dose of study treatment until end of study treatment (Day 1 to week 12) plus 8 weeks post-treatment follow-up epoch (week 12 to week 20).
Groups:
- Omalizumab 300 mg: Participants received omalizumab 300 mg subcutaneously every 4 weeks during the 12 week treatment period.
- Omalizumab 150 mg: Participants received omalizumab 150 mg subcutaneously every 4 weeks during the 12 week treatment period.
Arm/Group | Omalizumab 300 mg | Omalizumab 150 mg | Placebo
All-Cause Mortality (participants affected / at risk) | 0/167 | 0/167 | 0/83
Serious Adverse Events (participants affected / at risk) | 5/167 | 5/167 | 3/83
Other Adverse Events (participants affected / at risk) | 84/167 | 79/167 | 43/83
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Omalizumab 300 mg (N=167) | Omalizumab 150 mg (N=167) | Placebo (N=83)
Vertigo positional (Ear and labyrinth disorders) | 1 | 0 | 0
Pelvic inflammatory disease (Infections and infestations) | 0 | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 0 | 0
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Meniscus injury (Injury, poisoning and procedural complications) | 0 | 0 | 1
Ectopic pregnancy (Pregnancy, puerperium and perinatal conditions) | 0 | 1 | 0
Pregnancy (Pregnancy, puerperium and perinatal conditions) | 1 | 1 | 0
Cervical dysplasia (Reproductive system and breast disorders) | 0 | 1 | 0
Rectocele (Reproductive system and breast disorders) | 0 | 1 | 0
Urticaria chronic (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Embolism venous (Vascular disorders) | 0 | 0 | 1
Hypertension (Vascular disorders) | 1 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Omalizumab 300 mg (N=167) | Omalizumab 150 mg (N=167) | Placebo (N=83)
Abdominal discomfort (Gastrointestinal disorders) | 0 | 4 | 2
Diarrhoea (Gastrointestinal disorders) | 2 | 4 | 1
Pyrexia (General disorders) | 5 | 4 | 1
Hepatic function abnormal (Hepatobiliary disorders) | 0 | 2 | 3
Herpes zoster (Infections and infestations) | 1 | 4 | 0
Influenza (Infections and infestations) | 7 | 7 | 1
Nasopharyngitis (Infections and infestations) | 7 | 8 | 7
Pharyngitis (Infections and infestations) | 1 | 4 | 3
Upper respiratory tract infection (Infections and infestations) | 36 | 25 | 12
Urinary tract infection (Infections and infestations) | 4 | 1 | 2
Alanine aminotransferase increased (Investigations) | 1 | 6 | 1
Blood creatine phosphokinase increased (Investigations) | 1 | 5 | 0
Blood glucose increased (Investigations) | 2 | 0 | 2
Blood uric acid increased (Investigations) | 5 | 5 | 4
Lymphocyte count increased (Investigations) | 0 | 0 | 2
Platelet count decreased (Investigations) | 0 | 2 | 2
Red blood cells urine positive (Investigations) | 0 | 2 | 2
Hyperuricaemia (Metabolism and nutrition disorders) | 4 | 3 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 6 | 4 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 2
Dizziness (Nervous system disorders) | 1 | 2 | 2
Headache (Nervous system disorders) | 4 | 4 | 0
Hypoaesthesia (Nervous system disorders) | 2 | 0 | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 11 | 3 | 2
Dry throat (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 4 | 1 | 3
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 4 | 2 | 1
Dermatitis (Skin and subcutaneous tissue disorders) | 2 | 1 | 3
Eczema (Skin and subcutaneous tissue disorders) | 5 | 4 | 1
Hypertension (Vascular disorders) | 4 | 2 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (ie, data from all sites) in the clinical trial.

DOCUMENTS (2):
  • Study Protocol (2016-08-10): https://cdn.clinicaltrials.gov/large-docs/97/NCT03328897/Prot_000.pdf
  • Statistical Analysis Plan (2019-11-11): https://cdn.clinicaltrials.gov/large-docs/97/NCT03328897/SAP_001.pdf